CLINICAL TRIAL: NCT03290521
Title: The Role of Intraperitoneal Irrigation and Lavage With Normal Saline for Reduction of Postoperative Pain After Laparoscopic Hysterectomy and Myomectomy: A Randomized Controlled Trial
Brief Title: Intraperitoneal Lavage for Reducing Pain in Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Roberto Angioli, Director, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAINLESS2812
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-02

CONDITIONS: Pain, Postoperative
Keywords: pain; laparoscopy; washing; intraperitoneal irrigation
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients will therefore be divided into two groups:
  A - Yes Washing (SL) B - No Washing (NL)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - Yes Washing (SL) (Experimental): In this group, the washing process is continued. In particular, 1000cc of laced ringer is instilled by changing the position of the patient in Trendelenburg and Anti-Trendelenburg so that the liquid contacts not only the internal surgical wounds but the whole wall of the abdominal cavity.
  Interventions: Procedure: intraperitoneal washing with saline solution
- B- No Washing (NL) (Experimental): No washing was performed before the end of surgery
  Interventions: Procedure: No washing

INTERVENTIONS:
Procedure: intraperitoneal washing with saline solution — intraperitoneal washing at the end of surgery
  Arms: A - Yes Washing (SL)
Procedure: No washing — no washing
  Arms: B- No Washing (NL)

SUMMARY:
The aim of the present study is to evaluate the role of intraperitoneal washing irrigation with saline solution at the end of laparoscopic hysterectomy or myomectomy in reducing perception of postoperative pain.

DETAILED DESCRIPTION:
Patients will be fully and accurately informed on the type of intervention and will sign a specific informed consent, in accordance with CBM standards, both for the intervention to which the patient will undergo both for the study in question.

Randomization will be performed through a randomized randomization table generated by a computer. Patients will therefore be divided into two groups:

A - Yes Washing (SL) B - No Washing (NL) Prior to surgery, hemoglobin and PCR values will be evaluated in the preoperative.

Prior to the incision, an antibiotic prophylaxis will be performed with cefazoline 2gr intravenously.

The intervention in both groups involves the periombelic cutaneous incision and the sub-umbilical band. Introduction of 10mm led trocar based on open technique. The introduction of optics and CO2 insufflation allows the macroscopic visualization of the endotominal organs. The investigators proceed with the introduction of 3 additional 3-lane trocar accessories in the left iliac fossa, right and overlaid iliac thorax. You will perform a hysterectomy possibly associated with annessiectomy or myomectomy according to the surgical indication. Careful hemostasis is carried out. In the SL group, the washing process is continued. In particular, 1000cc of laced ringer is instilled by changing the position of the patient in Trendelenburg and Anti-Trendelenburg so that the liquid contacts not only the internal surgical wounds but the whole wall of the abdominal cavity. The surgery ends with the closure of the band and the breasts cutaneous. The parameters measured during the operation are: operating time, amount of CO2 injected (L), pneumoperitoneal pressure (mmHg). The operator surgeon is always the same.

In the postoperative period, the following parameters will be evaluated: hemoglobin, white blood cells, PCR, body temperature, recovery of intestinal activity, administration of toradol, paracetamol and possible morphine and postoperative postoperative pain, palpation, cough. The latter is evaluated through tables using the VAS visual scale: patients report the subjective characteristics of perceived postoperative pain by attributing a value of 0 (no pain) to 10 (worse pain than I can imagine). It assesses the occurrence of any complications in post-operative, infection and fever, which may require the patient's exclusion from the study.

ELIGIBILITY:
Inclusion Criteria:

* all patients candidates tor hysterectomy, hysterectomy and annessiectomy, laparoscopic myomectomy;
* ECOG Performance Status between 0 and 1;
* ages between 18 and 70 years
* no present or previous systemic neoplastic disease
* signed informed consent to the operation and execution of the intraperitoneal wash procedure.

Exclusion Criteria:

* pregnancy,
* pre-existing coagulopathy, neurological or cognitive dysfunction,
* previous or recent pelvic flogosis,
* previous opioid intake for chronic pain,
* previous abdominal surgery,
* previous or current systemic neoplastic disease
* concomitant ovarian and cervical gynecological disease,
* intraoperative conversion from laparoscopy to laparotomy ,
* intraoperative complications,
* use of morphine in the postoperative period,
* ECOG Performance Status >1.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
pain | 17 months
  to evaluate the postoperative pain using VAS scale

SECONDARY OUTCOMES:
infections | 17 months
  postoperative infections

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Angioli, Principal Investigator — Campus Bio-Medico University
Locations (1):
- Ethics Committee, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
Use of intraperitoneal washing to reduce postoperative pain in laparoscopy